CLINICAL TRIAL: NCT06656104
Title: Impact of a Multi-infusion Strategy in Neonatology on the Rate of Central Line-associated Bloodstream Infections
Acronym: EDELVAISS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0812; 2024-A00830-47 (Other: ID-RCB)
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Infection
Keywords: neonatal infection; prematurity; catheter; parenteral; perfusion
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Reference period: The center used the routine strategy based on the usual catheters and infusion systems (reference strategy). The duration of this period depending to the randomization of the center (i.e. 4 months, 8 months or 12 months)
  Interventions: Device: Reference strategy
- Experimental period: At the end of the reference period, center will progressively switch to the new multi-infusion strategy (experimental strategy). The center used the Multiline Neo system to the routine strategy. The duration of this period depending to the randomization of the center (i.e. 12 months, 8 months or 4 months)
  Interventions: Device: Experimental strategy

INTERVENTIONS:
Device: Reference strategy — Routine strategy based on the usual catheters and infusion systems used during the reference period
  Groups: Reference period
Device: Experimental strategy — EDELVAISS multi-infusion strategy as routine strategy during the experimental period
  Groups: Experimental period

SUMMARY:
The management of premature infants hospitalized in neonatal units requires the simultaneous intravenous (IV) infusion of several drugs and parenteral nutrition solutions, when oral administration is impossible or unsuitable. IV administration requires the use of a central venous catheter and an infusion set that connects the catheter to the infusion fluid or drug. The use of multiple infusion devices exposes patients to central line-associated bloodstream infections (CLABSI), drug interactions, abnormal administration timing and repetition of procedures in close proximity to the infant.

Against this backdrop, DORAN INTERNATIONAL has developed the EDELVAISS multi-infusion strategy (Multiline Neo® and Escape Line® devices) adapted to neonatology. Given its characteristics, the benefits expected from the use of this strategy are: 1) to reduce the risk of microbial contamination and therefore the number of nosocomial infections 2) reduce exposure to antibiotics used in late sepsis 3) reduce the number of central line losses due to catheter obstruction 4) reduce dys-stimulating procedures in contact with the infant and 5) reduce staff stress.

A pilot study before (year 2019) and after (year 2020) was carried out in the tertiary care neonatal unit at Croix-Rousse hospital. The baseline CLABSI rate was slightly below the national level of the last French survey (12.4/1000 catheter days [95%CI:10.8;14.0]). In 322 very-low-birth-weight infants, the investigators showed a significant 88% reduction in the rate of catheter-related bacteremia, from 11.3 to 2.2 infections per 1,000 catheter-days after implementation of the EDELVAISS multi-infusion strategy.

Since this pilot study, the EDELVAISS multi-infusion strategy has been used routinely in the neonatology department for around 2,000 infants admitted to the neonatology department at Croix-Rousse hospital. The low CLABSI rate observed in 2020 was maintained over the following 2 years. Several tertiary care neonatology departments have implemented the EDELVAISS multi-infusion strategy (ten departments have already done so, and five are in the process of doing so). The three neonatal units that agreed to take part in the EDELVAISS study also wish to implement the EDELVAISS multi-infusion strategy.

The invetsigators hypothesize that the reduction in CLABSI rates observed in the neonatal unit at Croix-Rousse hospital during the pilot study will be found in other French neonatal units, whatever the initial practices and devices used in each center.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth ≤ 32 weeks
* Birthweight ≤ 1600 g
* Admitted in the first 3 days of life in the neonatal unit
* Hospitalized in the neonatal unit for at least 1 day
* Survived the first three days of life
* Requires the use of infusion sets for the administration of multiple drugs or solutions, whether or not they have the device in place
* Receipt of the non-opposition from parents or guardians

Exclusion Criteria:

* Opposition by parents or guardians
* Lethal or complicated malformation
* Chromosomal anomaly
* Participation of the infant in any other research that may interfere with the results of this study, in the judgment of the investigator

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at less than 32 weeks and with a birth weight of less than 1600 g, requiring the use of a multi-infusion strategy to administrate several drugs or solutions.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of central line associated bloodstream infections (CLABSI) in very preterm infants | Up to six months
  The primary endpoint is the number of infections per 1000 catheter-days

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de néonatologie Hôpital Femme Mère Enfant, Bron, France
  - Service Pédiatrie néonatale et réanimations CHU Montpellier, Montpellier, France
  - Service de néonatologie CHU de Strasbourg, Strasbourg, France